CLINICAL TRIAL: NCT05420467
Title: A Prospective, Open-label, Non-inferiority Study to Evaluate Injectable Albumin-bound Paclitaxel Versus Docetaxel for the Adjuvant Treatment of Breast Cancer
Brief Title: A Study for the Adjuvant Treatment of Breast Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0056
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; adjuvant therapy; Docetaxel; albumin paclitaxel; TCbHP; nPCbHP; ddEC-wnP; TC; nPC; EC-T
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Carboplatin; Trastuzumab; pertuzumab; Taxes; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- TCbHP (Active Comparator): HER2-positive breast cancer
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab
- nPCbHP (Experimental): HER2-positive breast cancer
  Interventions: Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Nab paclitaxel
- EC-T (Active Comparator): Luminal breast cancer (HER2-, more than 4 lymph node metastases), and triple negative breast cancer
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- ddEC-wnP (Experimental): Luminal breast cancer (HER2-, more than 4 lymph node metastases), and triple negative breast cancer
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Nab paclitaxel
- TC (Active Comparator): Luminal breast cancer (HER2-, with 1-3 lymph nodes)
  Interventions: Drug: Docetaxel; Drug: Cyclophosphamide
- nPC (Experimental): Luminal breast cancer (HER2-, with 1-3 lymph nodes)
  Interventions: Drug: Nab paclitaxel; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2, d1, q3w,6 cycles
  Arms: TC; TCbHP
Drug: Carboplatin — AUC 6, d1, q3w,6 cycles
  Arms: TCbHP; nPCbHP
Drug: Trastuzumab — starting dose 8 mg/kg, maintenance dose 6 mg/kg, d1, q3w,6 cycles
  Arms: TCbHP; nPCbHP
Drug: Pertuzumab — starting dose of 840 mg, maintenance dose of 420 mg, d1, q3w ,6 cycles
  Arms: TCbHP; nPCbHP
Drug: Nab paclitaxel — 220 mg/m2, d1, q3w,6 cycles
  Arms: nPC; nPCbHP
Drug: Epirubicin — 90 mg/m2, d1, q3w ,4 cycles ,followed by docetaxel
  Arms: EC-T
Drug: Cyclophosphamide — 600 mg/m2, d1, q3w × 4 cycles followed by docetaxel
  Arms: EC-T
Drug: Docetaxel — 100 mg/m2, d1, q3w × 4 cycles
  Arms: EC-T
Drug: Epirubicin — 90 mg/m2,d1, q2w × 4 cycles followed by nab-paclitaxel
  Arms: ddEC-wnP
Drug: Cyclophosphamide — 600 mg/m2, d1, q2w × 4 cycles followed by nab-paclitaxel
  Arms: ddEC-wnP
Drug: Nab paclitaxel — 125 mg/m2, d1,8,15, q3w× 4 cycles
  Arms: ddEC-wnP
Drug: Cyclophosphamide — 600 mg/m2, d1, q3w × 6 cycles
  Arms: TC; nPC

SUMMARY:
Studies on postoperative adjuvant albumin paclitaxel in domestic breast cancer patients are less reported, especially in large samples, and more studies focus more on the safety and tolerability of albumin paclitaxel use. Head-to-head studies of white violet and docetaxel are not supported by data at this time, but some studies have shown that docetaxel-induced long-term Other adverse effects such as myelosuppression, hepatotoxicity and hypersensitivity reactions can have a serious impact on quality of life. Therefore, this study aims to analyse the efficacy and safety of albumin paclitaxel and docetaxel in the adjuvant treatment of breast cancer in a large randomized controlled trial, and to further analyse the efficacy and safety of albumin paclitaxel in combination with chemotherapy for postoperative breast cancer in different subtypes of breast cancer patients, in order to obtain more realistic data and provide new treatment options for breast cancer patients.

DETAILED DESCRIPTION:
At present, the treatment of early-stage breast cancer is mainly surgical, supplemented by chemotherapy, endocrine therapy, radiotherapy, targeted therapy and other comprehensive treatment methods, through the use of a variety of comprehensive and individualized treatment plans led to a significant improvement in the quality of life and survival of breast cancer patients. Systematic adjuvant therapy after surgery is also gaining increasing attention, with a large number of randomized clinical trials worldwide . The effectiveness of adjuvant therapy in reducing the recurrence of breast cancer and improving survival has been demonstrated in a number of randomized clinical trials worldwide. Adjuvant therapy after surgery is recommended in NCCN guidelines, ESMO, St. Gallen and other guidelines or expert consensus.

The use of albumin paclitaxel in the postoperative adjuvant treatment of breast cancer has been reported overseas, and a phase II clinical study published in 2017 investigated the tolerability and feasibility of dose dense doxorubicin combined with cyclophosphamide followed by nab-paclitaxel (AC-nP) chemotherapy in patients with high-risk early-stage breast cancer in adjuvant treatment. The results suggested that this regimen was well tolerated, with an incidence of granular deficiency with fever 5 of 2%, suggesting the safety of weekly treatment with nab-paclitaxel.

Another study evaluated the safety of dose-dense AC-nP regimens in women with high-risk breast cancer. Enrolled patients received 4 cycles of AC (every 2 weeks) followed by nab-P (every 2 weeks). The most common eventual adverse reaction was peripheral neuropathy, although approximately 80% of patients were grade 1-2, and the patient's neuropathy gradually improved after the end of treatment. This suggests that in early breast cancer, the use of dose-dense AC followed by nab-P is feasible with predictable AEs .

In summary, studies on postoperative adjuvant albumin paclitaxel in domestic breast cancer patients are less reported, especially in large samples, and more studies focus more on the safety and tolerability of albumin paclitaxel use. Head-to-head studies of white violet and docetaxel are not supported by data at this time, but some studies have shown that docetaxel-induced long-term Other adverse effects such as myelosuppression, hepatotoxicity and hypersensitivity reactions can have a serious impact on quality of life. Therefore, this study aim to conduct a prospective, randomized, open-label, multi-center clinical study to analyse the efficacy and safety of albumin paclitaxel and docetaxel in the adjuvant treatment of breast cancer in a large randomized controlled trial, and to further analyse the efficacy and safety of albumin paclitaxel in combination with chemotherapy for postoperative breast cancer in different subtypes of breast cancer patients, in order to obtain more realistic data and provide new treatment options for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 years;
2. Histopathologically or cytologically confirmed breast cancer patients with the following characteristics:1. stage I to III breast cancer; 2. operable primary lesion with no evidence of distant metastasis (M0);
3. known hormone receptor status (estrogen receptor [ER], progesterone receptor [PR]) and HER2 status with known Ki67 expression levels; (ER/PR positive defined as stained cells >1%, HER2 positive defined as IHC 3+ or IHC 2+ with a positive FISH test);
4. Triple-negative breast cancer (TNBC): ER/PR negative, HER2 negative; tumor >2cm or lymph node metastasis with clear postoperative pathological evidence; Luminal breast cancer: ER>1%, HER2 negative, postoperative pathological evidence definite lymph node metastasis (different adjuvant chemotherapy regimens depending on whether the lymph nodes are N1 or N2-3); HER2-positive breast cancer: HER2-positive, regardless of ER/PR status; (the above classification determines enrollment and adjuvant therapy, and does not represent the corresponding molecular typing definition);
5. Patients who have undergone breast cancer resection and systemic intrathoracic lymph node dissection; surgical resection is R0 resection; patients who need postoperative adjuvant chemotherapy as judged by the investigator;
6. Start of adjuvant therapy within 21 days of the time of surgery is appropriate ;
7. ECOG physical fitness score of 0-1 with an expected survival of >6 months ;
8. Patients have not been treated with a paclitaxel regimen prior to enrolment ;
9. Adjuvant chemotherapy should not be performed concurrently with endocrine therapy drugs such as tamoxifen/aromatase inhibitors or postoperative radiotherapy;
10. Women of childbearing age must have taken reliable contraceptive measures, or performed a pregnancy test (serum or urine) within 7 days before enrollment, with a negative result, and be willing to use appropriate contraceptives during the trial and 8 weeks after the last dose of the trial drug;
11. Electrocardiogram (ECG) and echocardiography must confirm normal cardiac function within 3 months prior to randomization. Left ventricular ejection fraction (LVEF) must be ≥55% for patients receiving anthracycline-containing chemotherapy regimens and targeted therapy ;
12. Liver and kidney function: serum creatinine ≤1.5 times the upper limit of normal; AST and ALT ≤3 times the upper limit of normal; total bilirubin ≤1.5 times the upper limit of normal, or ≤2.5 times the upper limit of normal when the patient has Gilbert's syndrome ;
13. Bone marrow function: neutrophils≥1.5×109/L, platelets≥100×109/L, hemoglobin≥90g/L;
14. Able to comply with outpatient treatment, laboratory monitoring and necessary clinical visits during the study period;
15. Subjects have the ability to understand, agree and sign the Informed Consent Form (ICF) for the study prior to initiating any protocol-related procedures; subjects have the ability to express consent (if applicable).

Exclusion Criteria:

1. Advanced and/or inoperable patients with distant metastasis confirmed by imaging evidence or pathology;
2. Other malignant tumors have occurred in the past 5 years, except for skin cancers of cured cervical carcinoma in situ and non-melanoma;
3. Pregnant or breastfeeding women; patients with childbearing potential who are unwilling or unable to take effective contraceptive measures;
4. The molecular status of ER/PR and HER2 and Ki67 cannot be determined;
5. Patients with CNS metastases or > grade 1 peripheral neuropathy;
6. Severe cardiovascular disease: Grade II or higher myocardial ischaemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥ 470 ms); Grade III-IV cardiac insufficiency according to NYHA criteria, or cardiac ultrasound indicating a left ventricular ejection fraction (LVEF) of <50%;
7. Patients with hypertension that cannot be reduced to the normal range after antihypertensive medication (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg);
8. Received major surgical operations or suffered severe traumatic injury, fracture or ulcer within 4 weeks of enrollment;
9. Patients with severe myelosuppression at screening;
10. Patients with severe liver dysfunction (Child's Class III) or renal dysfunction at screening ;
11. Arterial/venous thrombotic events such as cardiovascular and cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction, myocardial infarction), deep vein thrombosis and pulmonary embolism, that occurred within 6 months before randomization;
12. Patients with hypersensitivity to any of the components of albumin paclitaxel, epirubicin, cyclophosphamide, docetaxel, trastuzumab, and pertuzumab;
13. Patients with psychiatric disorders;
14. Subjects who are participating in another clinical study or whose first dose was administered less than 4 weeks (or 5 half-lives of the study drug) from the end of the previous clinical study (last dose) ;
15. The investigator judges other situations that may affect the clinical research and the judgment of the research results and are not suitable for inclusion in the research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2413 (Estimated)
Dates: Start 2022-07-10 (Estimated); Primary Completion 2027-07-10 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
5-year DFS | 5-years
  5-year disease-free survival

OTHER OUTCOMES:
DMFS | 2 years
  distant metastasis-free survival
OS | 10 years
  overall survival
RFS | 2 years
  recurrence-free survival
Remission rate of neurotoxicity | 5 years
The incidence of other AEs | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho E, Wu Q, Rubinstein L, Linden H, Gralow J, Specht J, Gadi V, Ellis G. Adjuvant continuous metronomic adriamycin + cyclophosphamide followed by weekly nab-paclitaxel for high-risk early-stage breast cancer. Breast J. 2018 Jul;24(4):610-614. doi: 10.1111/tbj.13013. Epub 2018 Mar 13. PMID 29532546
- [Background] Robert N, Krekow L, Stokoe C, Clawson A, Iglesias J, O'Shaughnessy J. Adjuvant dose-dense doxorubicin plus cyclophosphamide followed by dose-dense nab-paclitaxel is safe in women with early-stage breast cancer: a pilot study. Breast Cancer Res Treat. 2011 Jan;125(1):115-20. doi: 10.1007/s10549-010-1187-2. Epub 2010 Oct 14. PMID 20945091